CLINICAL TRIAL: NCT05684510
Title: Evaluation of Efficacy of Clear Aligners in Correction of Class II Malocclusion Using Intermaxillary Elastics: A Randomized Controlled
Brief Title: Treatment of Mild Class II Malocclusion in Adult Patients With Clear Aligners Versus Fixed Multibracket Therapy
Acronym: malocclusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hama University (Other)
Responsible Party: Principal Investigator, FADI JNAID, Syria-Hama University, Hama University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hama University -
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Malocclusion; Class II Malocclusion
MeSH Terms: conditions — Malocclusion; Overbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental : clear aligners with class II elastics technique (Experimental): clear aligners technique A group of patients in which participants will be undergo to clear aligners treatment with class II elastics ( clear aligners will be applied to the upper and lower arch, then a class II elastics 1\4 and 6,5 oz will be use from the precision-cut Hook on the maxillary aligner to the button of mandibular first molar
  Interventions: Device: clear aligners
- : traditional treatment Fixed appliances with class II elastics. (Experimental): A group of patients in which participants will be undergo to the fixed multibracket treatment (with slot size 0.022 × 0.028 and MBT prescription , after completing leveling and alignment , Elastics will be applied from the hooks of canines brackets to the hooks of lower first molar when the 0.019× 0.025-inch stainless steel archwires placed.
  Interventions: Device: traditional treatment Fixed appliances with class II elastics.

INTERVENTIONS:
Device: clear aligners — clear aligners will be applied to the upper and lower arch, then a class II elastics 1\4 and 6,5 oz will be use from the precision-cut Hook on the maxillary aligner to the button of mandibular first molar
  Arms: Experimental : clear aligners with class II elastics technique
Device: traditional treatment Fixed appliances with class II elastics. — Agroup of patients in which participants will be undergo to the fixed multibracket treatment (with slot size 0.022 × 0.028 and MBT prescription , after completing leveling and alignment , Elastics will be applied from the hooks of canines brackets to the hooks of lower first molar when the 0.019× 0.025-inch stainless steel archwires placed.
  Arms: : traditional treatment Fixed appliances with class II elastics.

SUMMARY:
Patient with class ii division 1 malocclusion who have mild increased overjet will be treated in this study. The efficacy of clear aligners in the treatment of Class II division 1 Malocclusion Using Intermaxillary Elastics will be assessed. The skeletal, dental and soft tissues changes resulted by this intervention will be studied and compared with the results of Traditional treatment with fixed appliances.

There are two group:

1. a group of patients in which participants will be undergo to the clear aligners with class ii elastics.
2. a group of patients in which participants will be undergo to the traditional fixed appliances with class ii elastics.

DETAILED DESCRIPTION:
Patient with class ii division 1 malocclusion who have mild increased overjet will be treated in this study. The efficacy of clear aligners in the treatment of Class II division 1 Malocclusion Using Intermaxillary Elastics will be assessed. The skeletal, dental and soft tissues changes resulted by this intervention will be studied and compared with the results of Traditional treatment with fixed appliances.

There are two group:

1. a group of patients in which participants will be undergo to the clear aligners with class ii elastics.
2. a group of patients in which participants will be undergo to the traditional fixed appliances with class ii elastics.

phase Intervention/treatment Condition or disease Not applicable Other: clear aligners Technique with class ii elastics. Other: fixed multibracket appliances with class ii elastics Malocclusion

Class ii Division 1 malocclusion

ELIGIBILITY:
Inclusion Criteria:

* - Patients with permanent occlusion at age 15-20 years.
* Patients with class II division I (half cusp or Less) with moderate overjet (2-4mm).
* Patients with normal or horizontal growth pattern.
* Mild crowding (_<2 mm) in maxillary and mandibular arch.
* Patient with satisfactory periodontal health and good oral hygiene
* No previous orthodontic treatment
* Comprehensive medical and dental history ruling out any systemic disease.

Exclusion Criteria:

* Patients with periodontal disease.
* Patients with vertical growth pattern.
* Patients with missing or extracted teeth except third molar.
* Patients with temporomandibular joint disorder.
* Patients with Skeletal open bite.
* Patients with poor oral and gingival health
* Patients with neuromuscular disorder.
* Patients with severe skeletal class II.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-08-25 (Estimated); Primary Completion 2026-11-11 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the SNA angle | : T0:1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 4-6 months in the exp. Group and 12 months in the control group
  This angle the represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in the SNB angle | : T0:1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved(expected to be within 4-6 months in the exp. Group and 12 months in the control group)
  This angle the represents the position of the lower jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in ANB angle | T0:1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 4-6 months in the exp. Group and 12 months in the control group)
  This angle the represents the spatial relationship between the upper and lower jaws in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in SN.POG angle | : T0: 1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 4-6 months in the exp. Group and 12 months in the control group)
  This angle the represents the position of the chin bone in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in the mandibular length [ | T0: 1day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 4-6 months in the exp. Group and 12 months in the control group)
  Amount of distance measured from the Co point to Gn point in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in SN.PP angle [ | T0: 1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved achieved (expected to be within 4-6 months in the exp. Group and 12 months in the control group)
  This angle the represents the amount and direction of rotation of the upper jaw in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in MP.SN angle | T0: 1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 4-6 months in the exp. Group and 12 months in the control group)
  This angle the represents the amount of backward rotation of the lower jaw in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
change in overjet | : T0: 1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 4-6 months in the exp. Group and 12 months in the control group)
  Represents The distance between the most anterior point on the lower incisor to the most anterior point on the upper incisor in the cephalometric analysis.
change in overbite | T0: 1 day before the beginning of treatment . T1: when a normal overjet and canines class I relationships achieved (expected to be within 4-6 months in the exp. Group and 12 months in the control group)
  Amount of coverage the upper incisor to lower incisor in the vertical plane in the cephalometric analysis.

CONTACTS AND LOCATIONS:
Overall Officials: FATIMA NASHTR, MSc, Principal Investigator — Hama University; Rabab AlSabbag, Professor, Study Director — Hama University
Locations (1):
- Hama University, Hama, Hama Governorate, Syria

IPD SHARING:
Plan to Share IPD: No